CLINICAL TRIAL: NCT02574832
Title: Determination of ED90 of Intrathecal Lidocaine for Adequate Anesthesia for Elective Cervical Cerclage Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: planned surgical procedures decreased
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Paloma Toledo, Assistant Professor in Anesthesiology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU0020134
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy; Surgery; Pain
Keywords: Pain; Surgery; Pregnancy; Anesthesia
MeSH Terms: conditions — Pain | interventions — Lidocaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Lidocaine Administration (Experimental): Spinal anesthesia will be induced with isobaric 2% lidocaine and 15 μg fentanyl.
  The study lidocaine dose will be determined using a 9:1 biased-coin sequential allocation method. For the first participant, the starting dose will be 32 mg of 2% isobaric lidocaine (1.6 mL). If the lidocaine dose provides an unsatisfactory anesthetic, the case will be categorized as a failure. After a failed case, the next participant will receive a lidocaine dose increased by 4 mg. If the lidocaine dose provides satisfactory anesthesia, the next participant's lidocaine dose will determined by a biased allocation method with a 90% chance of maintaining the dose and a 10% chance of decreasing the dose by 4 mg.
  Interventions: Drug: Lidocaine Administration

INTERVENTIONS:
Drug: Lidocaine Administration — The lidocaine dose will be determined using a 9:1 biased-coin sequential allocation method. For the first participant, the starting dose will be 32 mg of 2% isobaric lidocaine (1.6 mL). Two outcomes will be possible: satisfactory or unsatisfactory anesthesia.
  Other Names: Lidocaine 2 % plus 15 μg fentanyl

SUMMARY:
Cervical incompetence complicates approximately 1 in 500 pregnancies . Those women with cervical incompetence are at risk for second trimester spontaneous abortion and preterm labor. Cervical cerclage reduces these risks but must be performed under general or neuraxial anesthesia. Some anesthesiologists prefer neuraxial anesthesia, as it reduces fetal exposure to medications and avoids the risks associated with loss of maternal airway reflexes under general anesthesia. Spinal anesthesia, in particular, has the added advantage of being technically simple while still providing a rapid, dense sensory block. For cerclage placement, patients require a sensory block from the T10 to S4 dermatome in order to cover sensation from the cervix as well as the vagina and perineum. Patients presenting for cerclage under spinal anesthesia pose a dosing challenge given the physiologic changes associated with pregnancy. As women progress with their pregnancy, they require lower doses of intrathecal local anesthetic to achieve similar block level. Multiple studies have demonstrated that these changes start during the second trimester. Inadequate sensory coverage with a spinal anesthetic typically necessitates conversion to general anesthesia, causing additional time wasted and added risk to the patient and fetus. Anecdotally, this is the reason why some anesthesiologists choose general anesthesia for patients undergoing cerclage over a spinal anesthetic. As there is currently no literature determining the correct dosage for these patients, we propose a dose-response study to determine the ED90 of intrathecal lidocaine for adequate anesthesia for elective cervical cerclage placement.The findings of this study will help determine the minimum dose of intrathecal lidocaine necessary to provide adequate spinal anesthesia for cervical cerclage for 90% of women. This will help decrease the frequency of inadequate anesthesia for cervical cerclage.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is at least 18 years old
* ASA physical class I or II
* BMI <40 kg/m2,
* Presents for elective cervical cerclage during their first or second trimester of pregnancy will be eligible to participate.

Exclusion Criteria:

* Any patient who is not a candidate for neuraxial anesthesia (including coagulopathy,
* Local skin infection, uncorrected hypovolemia)
* Allergy to lidocaine or fentanyl
* Chronic opioid user
* History of failed neuraxial anesthesia or analgesia,
* Had prior spine surgery
* Can not assume a sitting position for spinal anesthesia due to risk of amniotic membrane rupture

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Toledo, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ioscovich A, Popov A, Gimelfarb Y, Gozal Y, Orbach-Zinger S, Shapiro J, Ginosar Y. Anesthetic management of prophylactic cervical cerclage: a retrospective multicenter cohort study. Arch Gynecol Obstet. 2015 Mar;291(3):509-12. doi: 10.1007/s00404-014-3391-5. Epub 2014 Aug 8. PMID 25103960
- [Background] Hirabayashi Y, Shimizu R, Saitoh K, Fukuda H. Spread of subarachnoid hyperbaric amethocaine in pregnant women. Br J Anaesth. 1995 Apr;74(4):384-6. doi: 10.1093/bja/74.4.384. PMID 7734254
- [Background] Lee GY, Kim CH, Chung RK, Han JI, Kim DY. Spread of subarachnoid sensory block with hyperbaric bupivacaine in second trimester of pregnancy. J Clin Anesth. 2009 Nov;21(7):482-5. doi: 10.1016/j.jclinane.2008.12.018. PMID 20006255
- [Background] Lee MH, Son HJ, Lee SH, Lee JH, Chung MH, Choi YR, Choi EM. Comparison of spread of subarachnoid sensory block and incidence of hypotension in early and late second trimester of pregnancy. Korean J Anesthesiol. 2013 Oct;65(4):322-6. doi: 10.4097/kjae.2013.65.4.322. Epub 2013 Oct 24. PMID 24228145
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Choi PT, Galinski SE, Takeuchi L, Lucas S, Tamayo C, Jadad AR. PDPH is a common complication of neuraxial blockade in parturients: a meta-analysis of obstetrical studies. Can J Anaesth. 2003 May;50(5):460-9. doi: 10.1007/BF03021057. PMID 12734154

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Lidocaine Administration: Spinal anesthesia will be induced with isobaric 2% lidocaine and 15 μg fentanyl.
  The study lidocaine dose will be determined using a 9:1 biased-coin sequential allocation method. For the first participant, the starting dose will be 32 mg of 2% isobaric lidocaine (1.6 mL). If the lidocaine dose provides an unsatisfactory anesthetic, the case will be categorized as a failure. After a failed case, the next participant will receive a lidocaine dose increased by 4 mg. If the lidocaine dose provides satisfactory anesthesia, the next participant's lidocaine dose will determined by a biased allocation method with a 90% chance of maintaining the dose and a 10% chance of decreasing the dose by 4 mg.
  Lidocaine Administration: The lidocaine dose will be determined using a 9:1 biased-coin sequential allocation method. For the first participant, the starting dose will be 32 mg of 2% isobaric lidocaine (1.6 mL). Two outcomes will be possible: satisfactory or unsatisfactory anesthesia.
Period: Overall Study
Arm/Group | Spinal Lidocaine Administration
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Lidocaine Administration
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 34 [30 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: count of participants]
  United States | 2
Height [Mean (Full Range); unit: centimeters] | 163.5 [162 to 165]
Weight [Mean (Full Range); unit: Kilograms] | 54.1 [48.1 to 60.1]
Number of live births [Mean (Full Range); unit: Number of live births] | 1 [1 to 1]
Indication for cerclage [Count of Participants; unit: Participants]
  Cervical Incompetence | 1
  History of previous loss | 1
Baseline heart rate [Mean (Full Range); unit: Beats per minute] | 73 [65 to 82]
Baseline systolic blood pressure [Mean (Full Range); unit: millimeters of mercury] | 111.5 [107 to 116]
Baseline diastolic blood pressure [Mean (Full Range); unit: millimeters of mercury] | 60 [57 to 63]
Estimated Gestational Age [Mean (Full Range); unit: weeks] | 13.3 [12.6 to 14]
Number of times pregnant [Mean (Full Range); unit: Number of pregnancies] | 4 [3 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Time to T 10 Level
Description: Elapsed time in minutes to achieve T 10 level of anesthesia. Assessed by the anesthesia care provider using crushed ice. T 10 level is numbness up to the level of the belly button.
Time Frame: 20 minutes after drug administration
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Spinal Lidocaine Administration
Number analyzed (Participants) | 2
Minutes | 12.5 [9 to 16]

ADVERSE EVENTS:
Time Frame: 24 hours after cerclage
Arm/Group | Spinal Lidocaine Administration
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Study ended early because of procedure changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No